CLINICAL TRIAL: NCT03738098
Title: NYCKidSeq: Incorporating Genomics Into Clinical Care of Diverse NYC Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Albert Einstein College of Medicine (Other); New York Genome Center (Other); National Human Genome Research Institute (NHGRI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Eimear Kenny, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 16-1731; U01HG009610 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Genetic Diseases, Inborn; Genetic Predisposition to Disease
Keywords: Whole Genome Sequencing; Genetic Counseling; Hereditary Childhood Disease; Genomic Medicine
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The overall design is a Randomized Controlled Trial (RCT), evaluating the use of GUÍA to facilitate the return of WGS genomic results and comparing it to return of results using routine genetic counseling. The RCT will occur in the context of the performing WGS and TGP for diagnostic purposes in 1,130 children in an effort to assess clinical utility. Children and young adults with specific disorders will be recruited from MS and EM. In the Traditional GC group, participants will receive traditional genetic counseling for the Baseline and Return of Results (ROR1) visits. In the GUÍA group, they will receive traditional GC for the Baseline visit, and traditional GC plus GUÍA for the ROR1 visit (see arm descriptions below). Based on the subjects' randomization, they will be scheduled to see a specific genetic counselor, as the genetic counselors will be assigned to a specific arm and will remain in that arm for the duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Genetic Counseling (Active Comparator): Standard of care genetic counseling session
  Interventions: Behavioral: Standard of Care
- GUÍA (Experimental): Standard of care genetic counseling session with Genomic Understanding, Information and Awareness (GUÍA).
  Interventions: Behavioral: Standard of Care; Behavioral: GUÍA

INTERVENTIONS:
Behavioral: Standard of Care — Participants will receive traditional genetic counseling (GC) for the Baseline and Return of Results (ROR1) visits.
  Other Names: Traditional Genetic Counseling
Behavioral: GUÍA — GUÍA for the ROR1 visit.
  Other Names: Communication Tool; Genomic Understanding, Information and Awareness
  Arms: GUÍA

SUMMARY:
The NYCKidSeq program will significantly advance the implementation of genomic medicine, particularly for children, young adults and their families in Harlem and the Bronx. The study will assess the clinical utility of genomic medicine in three broad areas of pediatric disorders, while engaging a range of providers and community advisors to overcome the well-documented barriers to inclusion of underserved and underrepresented populations in genomic research. The study will also include testing, analyzing, and implementing a novel communication tool, Genomic Understanding, Information and Awareness (GUÍA), to facilitate the return of genomic test results. The use of GUÍA will enhance the understanding of these genomic testing results by families, patients, and care providers at all levels of expertise, in two health systems. Healthcare system leadership will be engaged to provide insights into their readiness for genomic implementation. Overall, the NYCKidSeq program will inform the genomics and clinical communities about how to implement genomic medicine in a diverse population in a clinically useful, technologically savvy, culturally sensitive, and ethically sound manner.

DETAILED DESCRIPTION:
NYCKidSeq is a research study using a randomized controlled trial (RCT) design to compare the use of GUÍA in a traditional genetic counseling return of results session to facilitate the return of genomic results compared to a traditional return of results counseling session. GUÍA will be an enhanced, personalized electronic version focused on helping patients understand their own genomic results. The researchers will also evaluate the clinical utility of whole genome sequencing (WGS) compared to targeted gene panels (TGP) in children with suspected genetic etiology of their neurologic disorders, primary immunodeficiencies, and cardiovascular disorders with the goal of detecting the mutated gene(s) responsible for their disorder.

1100 referred children Mount Sinai and Albert Einstein College of Medicine/Montefiore Hospital (Einstein/Montefiore) will be enrolled and randomized to either traditional genetic counseling (standard of care) or traditional genetic counseling plus GUÍA. The researchers will assess parents' perceived and subjective understanding of results as well as their adherence to follow-up recommendation (primary and secondary outcomes) through the use of parental surveys at three time points. The RCT will occur in the context of performing WGS and TGP for diagnostic purposes in 1,130 children.

Participants will have three study visits (Baseline, ROR1, and ROR2) over a nine-month period. At the baseline visit, families will receive pre-test counseling and will complete a survey. Blood will be collected from all study participants and from each biological parent (if available) to assist with interpretation of genomic results. Samples will undergo WGS and TGP. Approximately three months later, results will be returned and explained via one of the two study arms - traditional genetic counseling versus genetic counseling with GUÍA, and parents will be asked to complete the ROR1 survey. Six months later, they will be asked to complete the ROR2 survey. The length of a subject's participation will be a minimum of nine months to a maximum of 27 months, depending on the time of study entry; participation after the initial nine months will consist solely of chart and data review. Over the initial 9-month period the investigators are studying the experiences and understanding of parents of children who receive sequencing to help understand how best to implement genomic medicine in a diverse population.

GUÍA will be an enhanced, personalized electronic version of a flip chart, which is the type of tool most commonly used in routine genetic counseling. In the third year of the study, the study team anticipates to have the tool integrated into EPIC. There are no tools yet focused on this complex information, specifically on helping patients understand their own genomic results.

ELIGIBILITY:
Inclusion Criteria:

* Infants, children and young adults up to and including 21 years of age; young adults (18-21) who are cognitively intact may participate in this study, but their parent(s) or legal guardian(s) must also agree to participate
* English- or Spanish-speaking parent or legal guardian capable of providing informed consent, participating in surveys, and able to see GUIA;
* Currently undiagnosed, likely genetic* cause of neurologic, immunologic, or cardiac disorders (*as determined by disorder-specific criteria in Section IIIc. and phenotype checklist Appendix w.)
* Followed by a physician in the MS or EM systems;
* Willing and able to return for each study visit (not moving out of the area within nine months)
* If targeted gene panels and/or whole exome sequencing were previously done, results must have been returned at least three months before enrollment;
* If targeted gene panels and/or whole exome sequencing were previously done, results must have been negative, or identified only one variant in a potentially causative autosomal recessive gene, and
* If the parents received genetic counseling about this child, themselves, or a family member, the last genetic counseling session must have been at least three months before enrollment (*if testing was within 6-months their recruitment will be held until they 3-months or after)
* If patients have undergone karyotyping alone, we do not have to wait 3 months prior to inclusion.

Exclusion Criteria:

* The referred child is currently participating in a different genetic sequencing study, that includes genetic counseling and/or return of results before the participant's ROR2 visit.
* The referred child has a known or likely molecular genetic diagnosis for their neurologic, immunologic, or cardiac disorder.
* The referred child has had a bone-marrow transplant.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 650 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Perceived understanding of genomic testing results | 3 months
  Perceived understanding of genomic testing results. Scale from 1 (very little or none of it) to 5 (understood almost all or all of it) at 3 months
Perceived understanding of genomic testing results | 9 months
  Perceived understanding of genomic testing results. Scale from 1 (very little or none of it) to 5 (understood almost all or all of it) at 3 months
Perceived confidence explaining genomic testing results | 3 months
  Perceived confidence explaining child's genetic test results. Scale from 1 (completely confident) to 5 (not confident at all) at 3 months
Perceived confidence explaining genomic testing results | 9 months
  Perceived confidence explaining child's genetic test results. Scale from 1 (completely confident) to 5 (not confident at all) at 9 months

SECONDARY OUTCOMES:
Objective understanding of genomic testing results | 3 months
  Participants will answer yes, no, or not sure/don't remember at 3 months
Objective understanding of genomic testing results | 9 months
  Participants will answer yes, no, or not sure/don't remember at 9 months
Understanding of recommended medical follow up and actionability of genomic results | 3 months
  Participants will answer yes, no, or I don't know/don't remember/unsure
Adherence to medical follow up recommendations | 9 months
  Participants will answer yes, not yet but plan to; or no, and don't plan to; or don't know
Percent of participants with definitive or likely positive diagnoses | up to 27 months
  Diagnostic results assessed by percent of participants with definitive or likely positive diagnoses
Time to diagnosis of WGS and TGP | up to 27 months
  Time to diagnosis comparison of WGS and TGP
Concordance of WGS and TGP results | up to 27 months
  Percent of agreement between WGS and TGP testing results

CONTACTS AND LOCATIONS:
Overall Officials: Eimear Kenny, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Melissa Wasserstein, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Albert Einstein College of Medicine/Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suckiel SA, Kelly NR, Odgis JA, Gallagher KM, Sebastin M, Bonini KE, Marathe PN, Brown K, Di Biase M, Ramos MA, Rodriguez JE, Scarimbolo L, Insel BJ, Ferar KDM, Zinberg RE, Diaz GA, Greally JM, Abul-Husn NS, Bauman LJ, Gelb BD, Horowitz CR, Wasserstein MP, Kenny EE. The NYCKidSeq randomized controlled trial: Impact of GUIA digitally enhanced genetic results disclosure in diverse families. Am J Hum Genet. 2023 Dec 7;110(12):2029-2041. doi: 10.1016/j.ajhg.2023.10.016. Epub 2023 Nov 24. PMID 38006881
- [Result] Abul-Husn NS, Marathe PN, Kelly NR, Bonini KE, Sebastin M, Odgis JA, Abhyankar A, Brown K, Di Biase M, Gallagher KM, Guha S, Ioele N, Okur V, Ramos MA, Rodriguez JE, Rehman AU, Thomas-Wilson A, Edelmann L, Zinberg RE, Diaz GA, Greally JM, Jobanputra V, Suckiel SA, Horowitz CR, Wasserstein MP, Kenny EE, Gelb BD. Molecular diagnostic yield of genome sequencing versus targeted gene panel testing in racially and ethnically diverse pediatric patients. Genet Med. 2023 Sep;25(9):100880. doi: 10.1016/j.gim.2023.100880. Epub 2023 May 6. PMID 37158195
- [Derived] Suckiel SA, Kelly NR, Odgis JA, Gallagher KM, Sebastin M, Bonini KE, Marathe PN, Brown K, Di Biase M, Ramos MA, Rodriguez JE, Scarimbolo L, Insel BJ, Ferar KDM, Zinberg RE, Diaz GA, Greally JM, Abul-Husn NS, Bauman LJ, Gelb BD, Horowitz CR, Wasserstein MP, Kenny EE. The NYCKidSeq randomized controlled trial: Impact of GUIA digitally enhanced genetic counseling in racially and ethnically diverse families. medRxiv [Preprint]. 2023 Jul 7:2023.07.05.23292193. doi: 10.1101/2023.07.05.23292193. PMID 37461450
- [Derived] Odgis JA, Gallagher KM, Suckiel SA, Donohue KE, Ramos MA, Kelly NR, Bertier G, Blackburn C, Brown K, Fielding L, Lopez J, Aguiniga KL, Maria E, Rodriguez JE, Sebastin M, Teitelman N, Watnick D, Yelton NM, Abhyankar A, Abul-Husn NS, Baum A, Bauman LJ, Beal JC, Bloom T, Cunningham-Rundles C, Diaz GA, Dolan S, Ferket BS, Jobanputra V, Kovatch P, McDonald TV, McGoldrick PE, Rhodes R, Rinke ML, Robinson M, Rubinstein A, Shulman LH, Stolte C, Wolf SM, Yozawitz E, Zinberg RE, Greally JM, Gelb BD, Horowitz CR, Wasserstein MP, Kenny EE. The NYCKidSeq project: study protocol for a randomized controlled trial incorporating genomics into the clinical care of diverse New York City children. Trials. 2021 Jan 14;22(1):56. doi: 10.1186/s13063-020-04953-4. PMID 33446240
- See also: Clinical Sequencing Evidence-Generating Research (CSER) Website — https://www.genome.gov/27546194/clinical-sequencing-evidencegenerating-research-cser2/